CLINICAL TRIAL: NCT06122259
Title: Multidisciplinary Surveillance and Investigation of Febrile Illness in Guinea
Brief Title: Febrile Illness in Guinea
Acronym: MuSIFe
Status: Recruiting | Type: Observational
Sponsor: Centre National de Formation et de Recherche en Sante Rurale (Other Government)
Collaborators: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Principal Investigator, Karifa Kourouma, Principal Investigator, Centre National de Formation et de Recherche en Sante Rurale
Other Study IDs: IRB/RR/AC/041_1616/22_ITM; 139/CNERS/23 (Other: Comité National d'Ethique pour la Recherche en Santé, Guinea); IRB/RR/AC/041_1616/22 (Other: Institutional Review Board of the Institute of Tropical Medicine, Antwerp, Belgium)
Record Dates: First submitted 2023-11-01; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Febrile Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Days
Biospecimen Retention: Samples With DNA — A venous blood volume of up to 10.5 ml will be collected from all participants to meet needs for routine clinical laboratory analysis and monitoring as well as study related laboratory analysis and sample storage needs at inclusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To date, the underlying causes of community-acquired fever, particularly non-malarial fever, are insufficiently documented in Guinea. Moreover, diagnostic capacity is limited, leading to inadequate prescription of antibiotics and antimalarials, as well as substantial delay in outbreak recognition. Thus, the investigators undertook a prospective observational multi-centric cohort study of febrile patients presenting at the emergency and outpatient department of selected health centers, districts and regional hospitals in four ecologically distinct sentinel health districts in Guinea.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥2 months old
* Documented fever (axillary temperature >37.5°C) at presentation or fever reported within the prior 24 hours
* Availability for follow-up for 21 days
* Willingness and ability of the patient or culturally acceptable representative to give informed consent for participation in the study

Exclusion Criteria:

* History of hospitalization (for > 48 hours within the last 14 days) at any health facility

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Febrile patients presenting with documented fever (> 37.5°C, axillary temperature) or reporting fever within the prior 24 hours (≤37.5°C, axillary temperature) at the emergency or outpatient department of the selected health facilities.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pattern of symptoms and laboratory results at presentation and during follow-up | Day 0 and day 21
  Proportion will be estimated
Syndromic and/or etiologic diagnoses as established at day 21 | Day 0
  Proportion will be estimated
Pattern and duration of antibiotic use (and other treatments) | Day 0
  Proportion and mean or median will be estimated
Immediate or secondary hospital admissions and of secondary/unscheduled visits | Day 0 and day 21
  Proportion will be estimated
Participants alive (with or without symptoms) or dead at day 21. | Day 21
  Survival or mortality rate will be estimated

SECONDARY OUTCOMES:
White blood cells and C-reactive protein levels at baseline and association with syndromic/etiologic diagnoses and with patient outcome at day 21 | Day 0
  Mean or median level will be estimated
Association of seasonal, geographical, demographic, clinical and first-line laboratory variables (malaria RDT and smear, biochemistry) with presenting syndromes/main etiologies | Day 0
  OR or RR will be estimated as appropriate
Confirmed arboviral pathogens and identification of epidemiological/clinical/laboratory predictors | Day 0
  Proportions will be estimated
Cases fulfilling any of the case definitions of the 20 epidemic-prone infections under surveillance as compared to the final diagnosis and proportion of them timely reported to health authorities | Day 0
  Proportions will be estimated

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Bottieau, MD, MSc, PhD, Study Director — Institute of Tropical Medicine, Antwerp, Belgium
Locations (1):
- Centre National de Formation et de Recherche en Santé Rurale, Maférinya, Forécariah, Guinea

IPD SHARING:
Plan to Share IPD: Yes
This is under development and will be filled when finalized.
Supporting Information: Study Protocol
Time Frame: Yet to be finalized.
Access Criteria: Yet to be finalized. However, investigators are opened to collaborate on that data that will be generated.

REFERENCES:
- [Background] World health organization. The WHO AWaRe (Access, Watch, Reserve) antibiotic book. WHO. 2022. https://www.who.int/publications/i/item/9789240062382. Accessed 11 Dec 2022
- [Result] Crump JA, Kirk MD. Estimating the Burden of Febrile Illnesses. PLoS Negl Trop Dis. 2015 Dec 3;9(12):e0004040. doi: 10.1371/journal.pntd.0004040. eCollection 2015 Dec. No abstract available. PMID 26633014
- [Result] Roddy P, Dalrymple U, Jensen TO, Dittrich S, Rao VB, Pfeffer DA, Twohig KA, Roberts T, Bernal O, Guillen E. Quantifying the incidence of severe-febrile-illness hospital admissions in sub-Saharan Africa. PLoS One. 2019 Jul 25;14(7):e0220371. doi: 10.1371/journal.pone.0220371. eCollection 2019. PMID 31344116
- [Result] Carugati M, Zhang HL, Kilonzo KG, Maze MJ, Maro VP, Rubach MP, Crump JA. Predicting Mortality for Adolescent and Adult Patients with Fever in Resource-Limited Settings. Am J Trop Med Hyg. 2018 Nov;99(5):1246-1254. doi: 10.4269/ajtmh.17-0682. PMID 30226134
- [Result] Alegana VA, Maina J, Ouma PO, Macharia PM, Wright J, Atkinson PM, Okiro EA, Snow RW, Tatem AJ. National and sub-national variation in patterns of febrile case management in sub-Saharan Africa. Nat Commun. 2018 Nov 26;9(1):4994. doi: 10.1038/s41467-018-07536-9. PMID 30478314
- [Result] Maze MJ, Bassat Q, Feasey NA, Mandomando I, Musicha P, Crump JA. The epidemiology of febrile illness in sub-Saharan Africa: implications for diagnosis and management. Clin Microbiol Infect. 2018 Aug;24(8):808-814. doi: 10.1016/j.cmi.2018.02.011. Epub 2018 Feb 15. PMID 29454844
- [Result] Prasad N, Murdoch DR, Reyburn H, Crump JA. Etiology of Severe Febrile Illness in Low- and Middle-Income Countries: A Systematic Review. PLoS One. 2015 Jun 30;10(6):e0127962. doi: 10.1371/journal.pone.0127962. eCollection 2015. PMID 26126200
- [Result] Steketee RW, Choi M, Linn A, Florey L, Murphy M, Panjabi R. World Malaria Day 2021: Commemorating 15 Years of Contribution by the United States President's Malaria Initiative. Am J Trop Med Hyg. 2021 Apr 23;104(6):1955-1959. doi: 10.4269/ajtmh.21-0432. PMID 33891560
- [Result] Iroh Tam PY, Obaro SK, Storch G. Challenges in the Etiology and Diagnosis of Acute Febrile Illness in Children in Low- and Middle-Income Countries. J Pediatric Infect Dis Soc. 2016 Jun;5(2):190-205. doi: 10.1093/jpids/piw016. Epub 2016 Apr 7. PMID 27059657
- [Result] Boillat-Blanco N, Mbarack Z, Samaka J, Mlaganile T, Kazimoto T, Mamin A, Genton B, Kaiser L, D'Acremont V. Causes of fever in Tanzanian adults attending outpatient clinics: a prospective cohort study. Clin Microbiol Infect. 2021 Jun;27(6):913.e1-913.e7. doi: 10.1016/j.cmi.2020.08.031. Epub 2020 Sep 4. PMID 32896654
- [Result] D'Acremont V, Kilowoko M, Kyungu E, Philipina S, Sangu W, Kahama-Maro J, Lengeler C, Cherpillod P, Kaiser L, Genton B. Beyond malaria--causes of fever in outpatient Tanzanian children. N Engl J Med. 2014 Feb 27;370(9):809-17. doi: 10.1056/NEJMoa1214482. PMID 24571753
- [Result] Wang H, Zhao J, Xie N, Wang W, Qi R, Hao X, Liu Y, Sevalie S, Niu G, Zhang Y, Wu G, Lv X, Chen Y, Ye Y, Bi S, Moseray M, Cellessy S, Kalon K, Baika DI, Luo Q. A Prospective Study of Etiological Agents Among Febrile Patients in Sierra Leone. Infect Dis Ther. 2021 Sep;10(3):1645-1664. doi: 10.1007/s40121-021-00474-y. Epub 2021 Jun 26. PMID 34173960
- [Result] Muianga A, Pinto G, Massangaie M, Ali S, Oludele J, Tivane A, Falk KI, Lagerqvist N, Gudo ES. Antibodies Against Chikungunya in Northern Mozambique During Dengue Outbreak, 2014. Vector Borne Zoonotic Dis. 2018 Aug;18(8):445-449. doi: 10.1089/vbz.2017.2261. Epub 2018 May 7. PMID 29733254
- [Result] Ushijima Y, Abe H, Nguema Ondo G, Bikangui R, Massinga Loembe M, Zadeh VR, Essimengane JGE, Mbouna AVN, Bache EB, Agnandji ST, Lell B, Yasuda J. Surveillance of the major pathogenic arboviruses of public health concern in Gabon, Central Africa: increased risk of West Nile virus and dengue virus infections. BMC Infect Dis. 2021 Mar 17;21(1):265. doi: 10.1186/s12879-021-05960-9. PMID 33731022
- [Result] World Health Organization. Integrated Management of Childhood Illness (IMCI)_chart booklet. Geneva; 2014. Link: https://www.who.int/publications/m/item/integrated-management-of-childhood-illness---chart-booklet-(march-2014)
- [Result] Shao AF, Rambaud-Althaus C, Samaka J, Faustine AF, Perri-Moore S, Swai N, Kahama-Maro J, Mitchell M, Genton B, D'Acremont V. New Algorithm for Managing Childhood Illness Using Mobile Technology (ALMANACH): A Controlled Non-Inferiority Study on Clinical Outcome and Antibiotic Use in Tanzania. PLoS One. 2015 Jul 10;10(7):e0132316. doi: 10.1371/journal.pone.0132316. eCollection 2015. PMID 26161535
- [Result] Guillebaud J, Bernardson B, Randriambolamanantsoa TH, Randrianasolo L, Randriamampionona JL, Marino CA, Rasolofo V, Randrianarivelojosia M, Vigan-Womas I, Stivaktas V, Venter M, Piola P, Heraud JM. Study on causes of fever in primary healthcare center uncovers pathogens of public health concern in Madagascar. PLoS Negl Trop Dis. 2018 Jul 16;12(7):e0006642. doi: 10.1371/journal.pntd.0006642. eCollection 2018 Jul. PMID 30011274
- [Result] van Griensven J, Cnops L, De Weggheleire A, Declercq S, Bottieau E. Point-of-Care Biomarkers to Guide Antibiotic Prescription for Acute Febrile Illness in Sub-Saharan Africa: Promises and Caveats. Open Forum Infect Dis. 2020 Jun 30;7(8):ofaa260. doi: 10.1093/ofid/ofaa260. eCollection 2020 Aug. PMID 32818139
- [Result] Keitel K, D'Acremont V. Electronic clinical decision algorithms for the integrated primary care management of febrile children in low-resource settings: review of existing tools. Clin Microbiol Infect. 2018 Aug;24(8):845-855. doi: 10.1016/j.cmi.2018.04.014. Epub 2018 Apr 21. PMID 29684634